CLINICAL TRIAL: NCT00980460
Title: Treatment of Children With All Stages of Hepatoblastoma With Temsirolimus (NSC#683864) Added to High Risk Stratum Treatment
Brief Title: Risk-Based Therapy in Treating Younger Patients With Newly Diagnosed Liver Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01975; NCI-2011-01975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AHEP0731; 10-00098; COG-AHEP0731; CDR0000654889; AHEP0731 (Other: Children's Oncology Group); AHEP0731 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH); NCT02265692 (obsolete NCT alias)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-06

CONDITIONS: PRETEXT I Hepatoblastoma; PRETEXT II Hepatoblastoma; PRETEXT III Hepatoblastoma; PRETEXT IV Hepatoblastoma
MeSH Terms: interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Dexrazoxane; Razoxane; Doxorubicin; Fluorouracil; dehydroftorafur; Irinotecan; Liver Transplantation; temsirolimus; Sirolimus; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- High-risk group (regimen H) (Experimental): Patients receive up front VIT chemotherapy comprising vincristine sulfate IV over 1 minute on days 1 and 8 and irinotecan hydrochloride IV over 90 minutes on days 1-5, and temsirolimus IV over 30 minutes on days 1 and 8. Treatment with VIT repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with disease response then receive 6 courses of C5VD with 4 courses of VIT in between each 2-course block. Patients with no disease response receive 6 courses of C5VD in the absence of disease progression or unacceptable toxicity. Patients undergo tumor resection or liver transplant after course 4 of C5VD followed by 2 courses of adjuvant C5VD. Patients may also receive dexrazoxane IV over 5-15 minutes on days 1-2 of courses 5 and 6.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Procedure: Liver Transplantation; Drug: Temsirolimus; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- High-risk group (regimen W) (Experimental): (regimen W replaced by regimen H as of Amendment 3B) Patients receive up front VI chemotherapy comprising vincristine sulfate IV on days 1 and 8 and irinotecan hydrochloride IV over 90 minutes on days 1-5. Treatment with VI repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with disease response then receive 6 courses of C5VD with 1 courses of VI in between each 2-course block. Patients with no disease response receive 6 courses of C5VD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Doxorubicin Hydrochloride; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- Intermediate-risk group (regimen F) (Experimental): Patients receive C5VD chemotherapy comprising cisplatin IV over 6 hours on day 1, fluorouracil IV over 2-4 minutes on day 2, vincristine sulfate IV over 1 minute on days 2, 9, and 16, and doxorubicin hydrochloride IV over 15 minutes on days 1-2. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo surgical resection after course 2 OR surgical resection or liver transplantation after course 4 of C5VD. Patients may also receive dexrazoxane IV over 5-15 minutes on days 1-2 of courses 5 and 6. (Closed to accrual as of 3/12/2012)
  Interventions: Drug: Cisplatin; Drug: Dexrazoxane; Drug: Doxorubicin Hydrochloride; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Procedure: Liver Transplantation; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- Low-risk group (regimen T) (Experimental): Patients undergo surgery and then receive adjuvant cisplatin IV over 6 hours on day 1, fluorouracil IV over 2-4 minutes on day 2, and vincristine sulfate IV over 1 minute on days 2, 9, and 16. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- Very low-risk group (Experimental): Patients undergo surgery and then receive no further treatment.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: High-risk group (regimen H); High-risk group (regimen W); Intermediate-risk group (regimen F); Low-risk group (regimen T)
Drug: Dexrazoxane — Given IV
  Other Names: 2, 6-Piperazinedione, 4,4'-propylenedi-, (P)- (8CI); 2,6-Piperazinedione, 4, 4'-(1-methyl-1,2-ethanediyl)bis-, (S)- (9CI); ADR 529; ADR-529; ADR529; ICRF 187; ICRF-187; ICRF187; Razoxane (+)-form; Soluble ICRF (L-isomer)
  Arms: Intermediate-risk group (regimen F)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: High-risk group (regimen H); High-risk group (regimen W); Intermediate-risk group (regimen F)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: High-risk group (regimen H); High-risk group (regimen W); Intermediate-risk group (regimen F); Low-risk group (regimen T)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
  Arms: High-risk group (regimen H); High-risk group (regimen W)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Liver Transplantation — Undergo liver transplant
  Other Names: Hepatic Transplantation; Liver Grafting; Liver Transplant; Transplantation of Liver
  Arms: High-risk group (regimen H); Intermediate-risk group (regimen F)
Drug: Temsirolimus — Given IV
  Other Names: CCI 779; CCI-779; CCI-779 Rapamycin Analog; CCI779; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: High-risk group (regimen H)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: High-risk group (regimen H); High-risk group (regimen W); Intermediate-risk group (regimen F); Low-risk group (regimen T)

SUMMARY:
This phase III trial studies the side effects and how well risk-based therapy works in treating younger patients with newly diagnosed liver cancer. Surgery, chemotherapy drugs (cancer fighting medicines), and when necessary, liver transplant, are the main current treatments for hepatoblastoma. The stage of the cancer is one factor used to decide the best treatment. Treating patients according to the risk group they are in may help get rid of the cancer, keep it from coming back, and decrease the side effects of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the event-free survival (EFS) in children with stage I (non-pure fetal histology [PFH], non-small cell undifferentiated [SCU]) and stage II (non-SCU) hepatoblastoma treated with surgical resection followed by 2 cycles of cisplatin, fluorouracil, and vincristine sulfate (C5V).

II. To determine the feasibility and toxicity of adding doxorubicin (doxorubicin hydrochloride) to the chemotherapy regimen of C5V for children with intermediate-risk hepatoblastoma.

III. To estimate the response rate to vincristine (vincristine sulfate), irinotecan (irinotecan hydrochloride), and temsirolimus in previously untreated children with high-risk, metastatic hepatoblastoma.

IV. To determine whether timely (between diagnosis and end of second cycle of chemotherapy) consultation with a treatment center with surgical expertise in major pediatric liver resection and transplant can be achieved in 70% of patients with potentially unresectable hepatoblastoma.

V. To foster the collection of tumor tissue and biologic samples to facilitate translational research and to provide data that may aid in risk-adapted approaches for subsequent clinical trials.

SECONDARY OBJECTIVES:

I. To estimate the EFS of patients with stage I PFH treated with surgery alone. II. To determine whether orthotopic liver transplantation (OLT) can be accomplished after successful referral and completion of 4 cycles of initial chemotherapy.

III. To estimate the 2-year EFS for patients once identified as candidates for possible OLT, the 2-year EFS for patients referred to a transplant center that are resected without OLT, and the 2-year EFS for patients referred to a transplant center who receive OLT.

IV. To register children with hepatoblastoma who receive OLT with PLUTO (Pediatric Liver Unresectable Tumor Observatory), an international cooperative registry for children transplanted for liver tumors.

V. To determine if pretreatment extent of disease (PRETEXT) grouping can predict tumor resectability.

VI. To monitor the concordance between institutional assessment of PRETEXT grouping and PRETEXT grouping as performed by expert panel review.

VII. To estimate the proportion of stage IV patients who have surgical resection of metastatic pulmonary lesions.

VIII. To determine the proportion and estimate the EFS of patients with potentially poor prognostic factors including alpha fetoprotein (AFP) < 100 ng/mL at diagnosis, microscopic positive surgical margins, surgical complications, multifocal tumors, microscopic vascular invasion, macrotrabecular histologic subtype, and SCU histologic subtype.

OUTLINE: Patients are assigned to 1 of 4 treatment groups according to risk group.

VERY LOW-RISK GROUP: Patients undergo surgery and receive no further treatment.

LOW-RISK GROUP: (regimen T) Patients undergo surgery and then receive adjuvant cisplatin intravenously (IV) over 6 hours on day 1, fluorouracil IV over 2-4 minutes on day 2, and vincristine sulfate IV over 1 minute on days 2, 9, and 16. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

INTERMEDIATE-RISK GROUP: (regimen F) (closed to accrual as of 3/12/2012) Patients receive C5VD chemotherapy comprising cisplatin IV over 6 hours on day 1, fluorouracil IV over 2-4 minutes on day 2, vincristine sulfate IV over 1 minute on days 2, 9, and 16, and doxorubicin hydrochloride IV over 15 minutes on days 1-2. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo surgical resection after course 2 OR surgical resection or liver transplantation after course 4 of C5VD. Patients may also receive dexrazoxane IV over 5-15 minutes on days 1-2 of courses 5 and 6.

HIGH-RISK GROUP: (regimen W) (regimen W replaced by regimen H as of Amendment 3B) Patients receive up front VI chemotherapy comprising vincristine sulfate IV on days 1 and 8 and irinotecan hydrochloride IV over 90 minutes on days 1-5. Treatment with VI repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with disease response then receive 6 courses of C5VD with 1 courses of VI in between each 2-course block. Patients with no disease response receive 6 courses of C5VD in the absence of disease progression or unacceptable toxicity.

HIGH-RISK GROUP: (regimen H) Patients receive up front VIT chemotherapy comprising vincristine sulfate IV over 1 minute on days 1 and 8 and irinotecan hydrochloride IV over 90 minutes on days 1-5, and temsirolimus IV over 30 minutes on days 1 and 8. Treatment with VIT repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients with disease response then receive 6 courses of C5VD with 4 courses of VIT in between each 2-course block. Patients with no disease response receive 6 courses of C5VD in the absence of disease progression or unacceptable toxicity. Patients undergo tumor resection or liver transplant after course 4 of C5VD followed by 2 courses of adjuvant C5VD. Patients may also receive dexrazoxane IV over 5-15 minutes on days 1-2 of courses 5 and 6.

After completion of study therapy, patients who receive chemotherapy are followed up periodically for at least 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with histologically-proven hepatoblastoma
* In emergency situations when a patient meets all other eligibility criteria and has had baseline required observations, but is too ill to undergo a biopsy safely, the patient may be enrolled on AHEP0731 without a biopsy

  * Clinical situations in which such emergent treatment may be indicated include, but are not limited to, the following circumstances:

    * Anatomic or mechanical compromise of critical organ function by tumor (e.g., respiratory distress/failure, abdominal compartment syndrome, urinary obstruction, etc)
    * Uncorrectable coagulopathy
  * For a patient to maintain eligibility for AHEP0731 when emergent treatment is given, the following must occur:

    * The patient must have a clinical diagnosis of hepatoblastoma, including an elevated alpha fetoprotein, and must meet all AHEP0731 eligibility criteria at the time of emergent treatment
    * Patient must be enrolled on AHEP0731 prior to initiating protocol therapy; a patient will be ineligible if any chemotherapy is administered prior to AHEP0731 enrollment
    * If the patient receives AHEP0731 chemotherapy PRIOR to undergoing a diagnostic biopsy, pathologic review of material obtained in the future during either biopsy or surgical resection must either confirm the diagnosis of hepatoblastoma or not reveal another pathological diagnosis to be included in the analysis of the study aims
* Patients will be staged for risk classification and treatment at diagnosis using Children's Oncology Group (COG) staging guidelines
* At the time of study enrollment, the patient's treatment regimen must be identified; if the patient's primary tumor was resected prior to the day of enrollment and a blood specimen for the determination of serum alpha fetoprotein was not obtained prior to that surgery, the patient will be considered to have alpha fetoprotein of greater than 100 ng/mL for the purpose of treatment assignment; if tumor samples obtained prior to the date of enrollment were not sufficient to determine whether small cell undifferentiated (SCU) histology was present, treatment assignment will be made assuming SCU is not present in the tumor
* For patients with stage I or II disease, specimens for rapid central review have been submitted and the rapid central review diagnosis and staging must be available to be provided on the AHEP0731 eligibility case report form (CRF)
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients may have had surgical resection of some or all sites of hepatoblastoma prior to enrollment
* Organ function requirements are not required for enrolled patients who are stage I, PFH and will not be receiving chemotherapy
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 mg/dL
  * 6 months to < 1 year: 0.5 mg/dL
  * 1 to < 2 years: 0.6 mg/dL
  * 2 to < 6 years: 0.8 mg/dL
  * 6 to < 10 years: 1 mg/dL
  * 10 to < 13 years: 1.2 mg/dL
  * 13 to < 16 years: 1.5 mg/dL (male) or 1.4 mg/dL (female)
  * >= 16 years: 1.7 mg/dL (male) or 1.4 mg/dL (female)
* Total bilirubin < 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 10 x ULN for age
* Absolute neutrophil count (ANC) > 750/uL
* Platelet count > 75,000/uL
* Shortening fraction >= 27% by echocardiogram
* Ejection fraction >= 47% by radionuclide angiogram (multi gated acquisition scan [MUGA]); Note: the echocardiogram (or MUGA) may be done within 28 days prior to enrollment
* Serum triglyceride level =< 300 mg/dL (=< 3.42 mmol/L)
* Serum cholesterol level =< 300 mg/dL (7.75 mmol/L)
* Random or fasting blood glucose within the upper normal limits for age; if the initial blood glucose is a random sample that is outside of the normal limits, then a follow-up fasting blood glucose can be obtained and must be within the upper normal limits for age
* Normal pulmonary function tests (including diffusing capacity of the lungs for carbon monoxide [DLCO]) if there is clinical indication for determination (e.g. dyspnea at rest, known requirement for supplemental oxygen); Note: for patients who do not have respiratory symptoms or requirement for supplemental oxygen, pulmonary function tests (PFTs) are NOT required
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and if seizures are well controlled
* Prothrombin time (PT) < 1.2 x ULN
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with stage I or II disease who do not have specimens submitted for rapid central pathology review by day 14 after initial surgical resection
* Patients that have been previously treated with chemotherapy for hepatoblastoma or other hepatoblastoma-directed therapy (e.g., radiation therapy, biologic agents, local therapy [embolization, radiofrequency ablation, laser]) are not eligible
* Patients who have received any prior chemotherapy are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anticancer agents are not eligible
* Patients who have previously received a solid organ transplant are not eligible
* Patients who have an uncontrolled infection are not eligible
* Females who are pregnant or breast feeding are not eligible for this study
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Males and females of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method
* Patients receiving corticosteroids are not eligible; patients must have been off corticosteroids for 7 days prior to start of chemotherapy
* Patients who are currently receiving enzyme inducing anticonvulsants are not eligible
* Patients must not be receiving any of the following potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers or inhibitors: erythromycin, clarithromycin, azithromycin, ketoconazole, itraconazole, voriconazole, posaconazole, grapefruit juice or St. John's wort
* Patients who are currently receiving therapeutic anticoagulants (including aspirin, low molecular weight heparin, warfarin and others) are not eligible
* Patients who are currently receiving angiotensin-converting enzymes (ACE) inhibitors are not eligible
* Patients must not have had major surgery within 6 weeks prior to enrollment on the high risk stratum; patients with history of recent minor surgical procedures (vascular catheter placement, bone marrow evaluation, laparoscopic surgery, liver tumor biopsy) will be eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Actual)
Dates: Start 2009-09-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M Katzenstein, Principal Investigator — Children's Oncology Group
Locations (209):
- United States (184):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Instituto De Oncologia Pediatrica, São Paulo, Brazil
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Japan (6):
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kagoshima University Medical Dental Hospital, Kagoshima, Kagoshima-ken
  - Shizuoka Cancer Center, Shizuoka, Suntou
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - National Cancer Center Hospital, Tokyo
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Thompson PA, Malogolowkin MH, Furman WL, Piao J, Krailo MD, Chung N, Brock L, Towbin AJ, McCarville EB, Finegold MJ, Ranganathan S, Dunn SP, Langham MR, McGahren ED, Tiao GM, Weldon CB, O'Neill AF, Rodriguez-Galindo C, Meyers RL, Katzenstein HM. Vincristine/irinotecan/temsirolimus upfront window treatment of high-risk hepatoblastoma: A report from the Children's Oncology Group AHEP0731 Study Committee. Pediatr Blood Cancer. 2023 Jul;70(7):e30365. doi: 10.1002/pbc.30365. Epub 2023 Apr 19. PMID 37073741
- [Derived] Trobaugh-Lotrario A, Katzenstein HM, Ranganathan S, Lopez-Terrada D, Krailo MD, Piao J, Chung N, Randazzo J, Malogolowkin MH, Furman WL, McCarville EB, Towbin AJ, Tiao GM, Dunn SP, Langham MR, McGahren ED, Feusner J, Rodriguez-Galindo C, Meyers RL, O'Neill AF, Finegold MJ. Small Cell Undifferentiated Histology Does Not Adversely Affect Outcome in Hepatoblastoma: A Report From the Children's Oncology Group (COG) AHEP0731 Study Committee. J Clin Oncol. 2022 Feb 10;40(5):459-467. doi: 10.1200/JCO.21.00803. Epub 2021 Dec 7. PMID 34874751
- [Derived] Katzenstein HM, Langham MR, Malogolowkin MH, Krailo MD, Towbin AJ, McCarville MB, Finegold MJ, Ranganathan S, Dunn S, McGahren ED, Tiao GM, O'Neill AF, Qayed M, Furman WL, Xia C, Rodriguez-Galindo C, Meyers RL. Minimal adjuvant chemotherapy for children with hepatoblastoma resected at diagnosis (AHEP0731): a Children's Oncology Group, multicentre, phase 3 trial. Lancet Oncol. 2019 May;20(5):719-727. doi: 10.1016/S1470-2045(18)30895-7. Epub 2019 Apr 8. PMID 30975630
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened for enrollment on 09/14/2009 and closed on 07/20/2018
Period: Overall Study
Arm/Group | Very Low-risk Group | Low-risk Group (Regimen T) | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen W) | High-risk Group (Regimen H)
Started | 8 | 51 | 105 | 32 | 40
Completed | 8 | 47 | 70 | 14 | 24
Not Completed | 0 | 4 | 35 | 18 | 16
Not completed — Death | 0 | 0 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 10 | 6 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 11 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Ineligible | 0 | 2 | 3 | 1 | 4
Not completed — Refusal of further therapy | 0 | 2 | 3 | 2 | 0
Not completed — No therapy within 42 days of resection | 0 | 0 | 3 | 1 | 0
Not completed — No transplant by protocol timepoints | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low-risk Group | Low-risk Group (Regimen T) | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen W) | High-risk Group (Regimen H) | Total
Number analyzed (Participants) | 8 | 51 | 105 | 32 | 40 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 51 | 105 | 32 | 40 | 236
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.5 (2.56) | 1.59 (1.71) | 1.42 (2.61) | 2.31 (2.4) | 2.75 (2.9) | 1.84 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 15 | 43 | 12 | 13 | 84
  Male | 7 | 36 | 62 | 20 | 27 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 13 | 27 | 10 | 16 | 67
  Not Hispanic or Latino | 7 | 35 | 73 | 22 | 23 | 160
  Unknown or Not Reported | 0 | 3 | 5 | 0 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 8 | 2 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 6 | 7 | 6 | 3 | 23
  White | 5 | 29 | 75 | 20 | 25 | 154
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 11 | 15 | 4 | 6 | 36
Region of Enrollment [Number; unit: participants]
  United States | 8 | 50 | 98 | 30 | 37 | 223
  Canada | 0 | 1 | 4 | 2 | 0 | 7
  Australia | 0 | 0 | 3 | 0 | 0 | 3
  Japan | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Estimated 5-year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients without an event are censored at last contact.
Time Frame: Time from patient enrollment to progression, treatment failure, death from any cause, diagnosis of a second malignant neoplasm, or last follow-up, assessed up to 5 years
Population: Only eligible patients are considered in the calculation of this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Very Low-risk Group | Low-risk Group (Regimen T) | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen W) | High-risk Group (Regimen H)
Number analyzed (Participants) | 8 | 49 | 102 | 31 | 36
Percent Probability | 100 [100 to 100] | 87.21 [73.67 to 94.06] | 87.03 [78.71 to 92.26] | 43.61 [25.79 to 60.16] | 46.38 [29.47 to 61.68]

2. Primary Outcome: Number of Cycles on Which Grade 3 or Higher Adverse Events Coded According to CTC AE Version 5 Were Observed
Description: All grade 3 or 4 or greater non-hematological toxicities. The frequency of each toxicity type will be quantified as the number of reporting periods on which the toxicity of the relevant grade is reported. This measure does not apply to patients enrolled in the VERY LOW RISK group.
Time Frame: During protocol therapy up to 1 year after enrollment
Population: All eligible patients except for patients in the very low-risk group. Regimen T includes 49 cycles, Regimen F includes 269 cycles, Regimen W includes 107 cycles and Regimen H includes 124 cycles.
Measure: Number; unit: Cycles
Units Other Than Participants: Cycles
Arm/Group | Low-risk Group (Regimen T) | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen W) | High-risk Group (Regimen H)
Number analyzed (Participants) | 51 | 105 | 32 | 40
Number analyzed (Cycles) | 49 | 269 | 107 | 124
Cycles
  Hearing impaired | 1 | 20 | 4 | 4
  Diarrhea | 4 | 15 | 15 | 15
  Enterocolitis | 1 | 0 | 0 | 1
  Nausea | 1 | 10 | 10 | 3
  Small intestinal obstruction | 1 | 1 | 0 | 0
  Vomiting | 2 | 24 | 13 | 5
  Abdominal distension | 0 | 1 | 3 | 0
  Abdominal pain | 0 | 10 | 9 | 6
  Colitis | 0 | 3 | 1 | 1
  Anal mucositis | 0 | 1 | 0 | 0
  Ascites | 0 | 1 | 0 | 0
  Malabsorption | 0 | 1 | 0 | 0
  Mucositis oral | 0 | 44 | 8 | 6
  Constipation | 0 | 2 | 1 | 0
  Dental caries | 0 | 1 | 0 | 0
  Typhlitis | 0 | 2 | 2 | 1
  Duodenal obstruction | 0 | 1 | 0 | 0
  Esophageal hemorrhage | 0 | 1 | 0 | 0
  Gastritis | 0 | 1 | 1 | 0
  Illeus | 0 | 3 | 4 | 0
  Oral pain | 0 | 4 | 1 | 0
  Small intestinal mucositis | 0 | 1 | 0 | 0
  Colonic hemorrhage | 0 | 0 | 1 | 0
  Dysphagia | 0 | 0 | 1 | 0
  Esophagitis | 0 | 0 | 1 | 0
  Gastroparesis | 0 | 0 | 1 | 0
  Gastric fistula | 0 | 0 | 0 | 1
  Gastrointestinal disorders - Other, specify | 0 | 0 | 0 | 1
  Obstruction gastric | 0 | 0 | 0 | 1
  Rectal mucositis | 0 | 0 | 0 | 1
  Fever | 1 | 9 | 1 | 9
  General disorders and administration site conditions - Other, specify | 0 | 1 | 0 | 0
  Pain | 0 | 6 | 1 | 4
  Multi-organ failure | 0 | 1 | 0 | 2
  Irritability | 0 | 0 | 0 | 1
  Infusion related reaction | 0 | 0 | 0 | 1
  Hypothermia | 0 | 0 | 0 | 1
  Catheter related infection | 1 | 8 | 1 | 0
  Infections and infestations - Other, specify | 4 | 38 | 27 | 9
  Mucosal infection | 1 | 0 | 1 | 0
  Otitis media | 1 | 0 | 1 | 0
  Urinary tract infection | 1 | 3 | 0 | 3
  Biliary tract infection | 0 | 1 | 0 | 0
  Abdominal infection | 0 | 1 | 0 | 0
  Bladder infection | 0 | 2 | 0 | 0
  Enterocolitis infectious | 0 | 8 | 4 | 5
  Duodenal infection | 0 | 1 | 0 | 0
  Upper respiratory infection | 0 | 4 | 2 | 2
  Eye infection | 0 | 1 | 0 | 0
  Wound infection | 0 | 1 | 0 | 0
  Sepsis | 0 | 5 | 0 | 3
  Lung infection | 0 | 2 | 0 | 1
  Peritoneal infection | 0 | 1 | 0 | 0
  Skin infection | 0 | 1 | 1 | 7
  Small intestine infection | 0 | 1 | 0 | 0
  Periorbital infection | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 1 | 28 | 9 | 6
  Aspartate aminotransferase increased | 1 | 37 | 10 | 19
  Activated partial thromboplastin time prolonged | 0 | 2 | 3 | 1
  Alkaline phosphatase increased | 0 | 1 | 0 | 1
  Blood bilirubin increased | 0 | 7 | 2 | 5
  Creatinine increased | 0 | 3 | 0 | 1
  GGT increased | 0 | 7 | 1 | 6
  Weight loss | 0 | 6 | 4 | 6
  Fibronogen decreased | 0 | 2 | 0 | 1
  Ejection fraction decreased | 0 | 1 | 0 | 1
  Investigations - Other, specify | 0 | 1 | 0 | 0
  White blood cell decreased | 0 | 0 | 1 | 0
  INR increased | 0 | 0 | 1 | 0
  CPK increased | 0 | 0 | 0 | 1
  Cholesterol high | 0 | 0 | 0 | 1
  Electrocardiogram QT corrected interval prolonged | 0 | 0 | 0 | 1
  Lipase increased | 0 | 0 | 0 | 1
  Serum amylase increased | 0 | 0 | 0 | 1
  Anorexia | 1 | 30 | 20 | 17
  Dehydration | 3 | 13 | 3 | 12
  Hyperglycemia | 2 | 15 | 5 | 10
  Hyperkalemia | 2 | 12 | 3 | 5
  Hypermagnesemia | 2 | 4 | 0 | 0
  Hypernatremia | 2 | 1 | 0 | 3
  Hypokalemia | 4 | 48 | 12 | 29
  Hyponatremia | 1 | 22 | 6 | 10
  Acidosis | 0 | 4 | 0 | 1
  Alkalosis | 0 | 1 | 0 | 3
  Hypocalcemia | 0 | 7 | 4 | 2
  Hypoalbuminemia | 0 | 3 | 3 | 1
  Hypomagnesemia | 0 | 11 | 3 | 2
  Hypophosphatemia | 0 | 21 | 7 | 19
  Tumor lysis syndrome | 0 | 2 | 0 | 0
  Hypercalcemia | 0 | 0 | 1 | 0
  Hypoglycemia | 0 | 0 | 1 | 1
  Hypertriglyceridemia | 0 | 0 | 0 | 4
  Metabolism and nutrition disorders - Other, specify | 0 | 0 | 0 | 1
  Peripheral sensory neuropathy | 2 | 5 | 2 | 1
  Oculomotor nerve disorder | 0 | 3 | 0 | 0
  Abducens nerve disorder | 0 | 1 | 2 | 0
  Peripheral motor neuropathy | 0 | 7 | 3 | 2
  Syncope | 0 | 1 | 0 | 0
  Dysphasia | 0 | 0 | 1 | 0
  Depressed level of consciousness | 0 | 0 | 0 | 1
  Seizure | 0 | 0 | 0 | 1
  Apnea | 1 | 0 | 0 | 0
  Atelectasis | 0 | 2 | 0 | 0
  Dyspnea | 0 | 2 | 1 | 3
  Bronchospasm | 0 | 1 | 0 | 0
  Hypoxia | 0 | 10 | 2 | 6
  Pleural effusion | 0 | 2 | 2 | 1
  Pulmonary edema | 0 | 1 | 0 | 0
  Stridor | 0 | 1 | 0 | 0
  Respiratory failure | 0 | 2 | 0 | 1
  Epistaxis | 0 | 0 | 2 | 1
  Wheezing | 0 | 0 | 0 | 1
  Hypertension | 3 | 6 | 2 | 4
  Hematoma | 0 | 1 | 1 | 0
  Hypotension | 0 | 3 | 3 | 5
  Vascular disorders - Other, specify | 0 | 2 | 1 | 0
  Thromboembolic event | 0 | 0 | 1 | 1
  Left ventricular systolic dysfunction | 0 | 1 | 1 | 0
  Cardiac arrest | 0 | 1 | 3 | 0
  Right ventricular dysfunction | 0 | 2 | 0 | 0
  Ventricular tachycardia | 0 | 1 | 0 | 0
  Cardiac disorders - Other, specify | 0 | 0 | 1 | 0
  Sinus tachycardia | 0 | 0 | 1 | 4
  Heart failure | 0 | 0 | 1 | 1
  Myocardial infarction | 0 | 0 | 1 | 0
  Biliary fistula | 0 | 1 | 0 | 0
  Hepatobiliary disorders - Other, specify | 0 | 1 | 0 | 1
  Hepatic hemorrhage | 0 | 2 | 1 | 1
  Portal vein thrombosis | 0 | 1 | 0 | 0
  Portal hypertension | 0 | 0 | 1 | 0
  Biliary anastomotic leak | 0 | 1 | 1 | 0
  Postoperative hemorrhage | 0 | 1 | 1 | 0
  Gastrointestinal anastomotic leak | 0 | 0 | 2 | 0
  Intraoperative hemorrhage | 0 | 0 | 0 | 1
  Arthralgia | 0 | 1 | 0 | 0
  Generalized muscle weakness | 0 | 2 | 0 | 0
  Back pain | 0 | 1 | 0 | 0
  Bone pain | 0 | 1 | 0 | 0
  Muscle weakness lower limb | 0 | 1 | 0 | 0
  Agitation | 0 | 4 | 1 | 0
  Hallucinations | 0 | 1 | 0 | 0
  Insomnia | 0 | 0 | 0 | 1
  Acute kidney injury | 0 | 9 | 0 | 0
  Renal and urinary disorders - Other, specify | 0 | 3 | 1 | 0
  Renal calculi | 0 | 1 | 0 | 0
  Proteinuria | 0 | 0 | 0 | 1
  Erythema multiforme | 0 | 1 | 0 | 0
  Skin and subcutaneous tissue disorders - Other, specify | 0 | 2 | 0 | 1
  Rash maculo-papular | 0 | 3 | 1 | 2
  Eye disorders - Other, specify | 0 | 1 | 0 | 0
  Surgical and medical procedures - Other, specify | 0 | 1 | 0 | 0
  Tumor pain | 0 | 0 | 1 | 0
  Allergic reaction | 0 | 0 | 0 | 2
  Anaphylaxis | 0 | 0 | 0 | 2
  Immune system disorders - Other, specify | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Deaths
Description: Number of patients who experience on-protocol-therapy death possibly, probably or likely related to systemic chemotherapy. This outcome measure applies to INTERMEDIATE RISK patients only.
Time Frame: During protocol therapy or within 30 days of the termination of protocol therapy up to 1 year after enrollment
Population: Only eligible patients are considered in the calculation of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate-risk Group (Regimen F)
Number analyzed (Participants) | 102
Participants | 1

4. Primary Outcome: Disease Status at the End of 2 Courses of Therapy
Description: RECIST v 1.1 and serum alphafetoprotein responses are evaluated separately. RECIST v 1.1 complete response (CR) is defined as disappearance of all target lesions and partial response (PR) is defined as reduction of at last 30% in the sum of the longest dimension of all target lesions (CR and PR measured by CT or MRI) between enrollment. Serum alphafetoprotein response is a decrease of at least 90% from the last serum alphafetoprotein measurement from the baseline prior to the start of chemotherapy to the end of cycle 2. This is calculated for HIGH RISK regimen W and HIGH RISK regimen H only.
Time Frame: First two cycles of therapy- up to 42 days after enrollment
Population: Thirty-two (32) patients were enrolled to Regiment W. Two were excluded from the analysis: (1)one was ineligible; and (2) one did not have an accurate report of initial AFP. Forty (40) patients were enrolled to Regiment H. Five were excluded from the analysis: (1)four were ineligible; and (2) one did not receive Temsirolimus.
Measure: Number; unit: participants
Arm/Group | High-risk Group (Regimen W) | High-risk Group (Regimen H)
Number analyzed (Participants) | 30 | 35
participants
  RECIST PR, no AFP response | 3 | 3
  AFP response, no RECIST response | 5 | 10
  RECIST response, AFP response | 6 | 4
  no AFP response, no RECIST response | 16 | 18

5. Secondary Outcome: Feasibility of Referral for Liver Transplantation
Description: A patient for whom referral is considered appropriate who receives a consultation after enrollment will be considered a success with respect to feasibility.
Time Frame: 3 cycles of therapy - up to 3 months after enrollment
Population: Only eligible patients with COG surgical stage III or IV disease and whose tumor is PRETEXT classified as PRETEXT 3-4 extensive multifocal; PRETEXT 3 +V; PRETEXT 3 +P; or PRETEXT 4 extensive multifocal are evaluated for feasibility of transplant referral.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen H)
Number analyzed (Participants) | 57 | 31
Participants | 37 | 16

ADVERSE EVENTS:
Time Frame: AEs and OAEs: Up to 6 months post-treatment planned as 18 months; All-Cause Mortality: up to 10 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Very Low-risk Group | Low-risk Group (Regimen T) | Intermediate-risk Group (Regimen F) | High-risk Group (Regimen W) | High-risk Group (Regimen H)
All-Cause Mortality (participants affected / at risk) | 0/8 | 3/49 | 7/102 | 11/31 | 13/36
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/49 | 3/102 | 2/31 | 1/36
Other Adverse Events (participants affected / at risk) | 0/8 | 24/49 | 91/102 | 27/31 | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Very Low-risk Group (N=8) | Low-risk Group (Regimen T) (N=49) | Intermediate-risk Group (Regimen F) (N=102) | High-risk Group (Regimen W) (N=31) | High-risk Group (Regimen H) (N=36)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Very Low-risk Group (N=8) | Low-risk Group (Regimen T) (N=49) | Intermediate-risk Group (Regimen F) (N=102) | High-risk Group (Regimen W) (N=31) | High-risk Group (Regimen H) (N=36)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 7 | 3 | 5
Abducens nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 2 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 5 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 3 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 21 | 7 | 6
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 2
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 19 | 9 | 11
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 26 | 7 | 16
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bladder infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 7 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 5 | 1 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
CPK increased (Investigations) | 0 | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 8 | 2 | 10
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 4 | 12 | 8 | 13
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Duodenal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 6 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 50 | 19 | 14
Fever (General disorders) | 0 | 1 | 8 | 0 | 11
Fibrinogen decreased (Investigations) | 0 | 0 | 2 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 6 | 1 | 5
Hallucinations (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 18 | 2 | 4
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 14 | 2 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 9 | 3 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 3 | 4 | 2 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 7 | 4 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4 | 37 | 7 | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 11 | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 15 | 4 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 18 | 6 | 13
Hypotension (Vascular disorders) | 0 | 0 | 1 | 2 | 4
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 1 | 6
Ileus (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 4 | 26 | 16 | 7
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 30 | 5 | 6
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 8 | 4 | 3
Neutrophil count decreased (Investigations) | 0 | 3 | 4 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 6 | 1 | 2
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 4 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 4 | 1 | 1
Peritoneal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 2
Rectal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 4 | 0 | 3
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 5
Small intestinal mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Small intestine infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 4 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 3
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 2 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 19 | 9 | 4
Weight loss (Investigations) | 0 | 0 | 4 | 3 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT00980460/Prot_SAP_000.pdf